CLINICAL TRIAL: NCT03357263
Title: Randomized, Single-Blind, Active Comparator-controlled Study to Evaluate the Safety and Immunological Efficacy of GC3114 in Healthy Adults.
Brief Title: A Study to Evaluate the Safety and Efficacy(Immunogenicity) of GC3114 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GC3114_P1
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC3114 (Experimental): Pre-filled syringe inj., 0.5ml, Once, IM
  Interventions: Biological: GC3114
- GCFLU Quadrivalent (Active Comparator): Pre-filled syringe inj., 0.5ml, Once, IM
  Interventions: Biological: GCFLU Quadrivalent

INTERVENTIONS:
Biological: GC3114 — High-dose Quadrivalent influenza vaccine
  Arms: GC3114
Biological: GCFLU Quadrivalent — Quadrivalent influenza vaccine
  Arms: GCFLU Quadrivalent

SUMMARY:
Healthy adults will be once administered GC3114A(High-dose Quadrivalent influenza vaccine) or GCFLU Quadrivalent Pre-filled syringe inj..

DETAILED DESCRIPTION:
Healthy adults will be once administered GC3114A(High-dose Quadrivalent influenza vaccine) or GCFLU Quadrivalent Pre-filled syringe inj.. Safety and immunological efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19-64 years old
* Informed consent form has been signed and dated
* Able to comply with the requirements of the study

Exclusion Criteria:

* Known systemic hypersensitive to eggs, chicken proteins, or any of the vaccine components
* Personal history of Guillain-Barre syndrome(GBS)
* Subjects with severe chronic disease who are considered by investigator to be ineligible for the study
* Subjects who received a vaccination within 28 days before enrollment or who are scheduled for another vaccination during the study
* Immunocompromised subjects with immunodeficiency disease or subjects receiving immunosuppressive or immunomodulating therapy
* Pregnant or lactating women

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Adverse Event | for 7 days from Day0/during study period
  Solicited/Unsolicited Adverse Event

SECONDARY OUTCOMES:
Percentage of participants achieving pre-defined Seroconversion Before and following vaccination | Day 0 and Day 21
  Seroconversion rate (SCR)
Percentage of participants achieving pre-defined Seroprotection Before and following vaccination | Day 0 and Day 21
  Seroprotection rate (SPR)
Geometric Mean Titer and Geometric Mean Titer Ratios of Antibodies to the Investigational Product Before and Following vaccination | Day 0 and Day 21
  Geometric Mean Titer(GMT), Geometric Mean Titer(GMT)

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo KIm, M.D, Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noh JY, Jang YS, Lee SN, Choi MJ, Yoon JG, Yu DH, Song JY, Cheong HJ, Kim WJ. Randomized, single-blind, active-controlled phase I clinical trial to evaluate the immunogenicity and safety of GC3114 (high-dose, quadrivalent influenza vaccine) in healthy adults. Vaccine. 2019 Aug 23;37(36):5171-5176. doi: 10.1016/j.vaccine.2019.07.076. Epub 2019 Jul 31. PMID 31377075